CLINICAL TRIAL: NCT03961529
Title: A Multicenter, Open-label, Uncontrolled, Long-term Trialto Demonstrate the Safety and Efficacy of 1% OPA-15406 Ointment in Adult Patients With Atopic Dermatitis and of 0.3% and 1% OPA-15406 Ointments in Pediatric Patients With Atopic Dermatitis (Phase 3 Trial)
Brief Title: Long-term Trial of OPA-15406 Ointment in Adult and Pediatric Patients With Atopic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 271-102-00006
Record Dates: First submitted 2019-04-26; First posted 2019-05-23 (Actual); Results first posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 0.3% OPA-15406 ointment (Experimental): Twice daily
  Interventions: Drug: 0.3% OPA-15406 ointment
- 1% OPA-15406 ointment (Experimental): Twice daily
  Interventions: Drug: 1% OPA-15406 ointment

INTERVENTIONS:
Drug: 0.3% OPA-15406 ointment — Twice daily
  Arms: 0.3% OPA-15406 ointment
Drug: 1% OPA-15406 ointment — Twice daily
  Arms: 1% OPA-15406 ointment

SUMMARY:
To demonstrate the safety of 1% OPA-15406 ointment in adult patients with AD and of 0.3% and 1% OPA-15406 ointments in pediatric patients with AD administered twice daily for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age: At least 2 years (at time of obtaining informed consent)
* Diagnosis of AD based on the Japanese Dermatological Association's criteria
* Atopic dermatitis affecting ≥5% of body surface area (BSA, excluding scalp) at the screening and baseline examinations

Exclusion Criteria:

- Subjects who have an AD or contact dermatitis flare-up defined as a rapid intensification of AD, within 28 days prior to the baseline examination

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2019-05-14 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Sato, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Shirao clinic of pediatrics and pediatric allergy, Hiroshima, Japan

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

REFERENCES:
- [Derived] Saeki H, Imamura T, Yokota D, Tsubouchi H. Difamilast Ointment in Japanese Adult and Pediatric Patients with Atopic Dermatitis: A Phase III, Long-Term, Open-Label Study. Dermatol Ther (Heidelb). 2022 Jul;12(7):1589-1601. doi: 10.1007/s13555-022-00751-9. Epub 2022 Jun 18. PMID 35716332

RESULTS

PARTICIPANT FLOW:
Groups:
- Adult: 1% OPA-15406 Ointment; Pediatric: 0.3% OPA-15406 Ointment; Pediatric: 1% OPA-15406 Ointment: Twice daily
Period: Overall Study
Arm/Group | Adult: 1% OPA-15406 Ointment | Pediatric: 0.3% OPA-15406 Ointment | Pediatric: 1% OPA-15406 Ointment
Started | 166 | 144 | 56
Completed | 124 | 127 | 51
Not Completed | 42 | 17 | 5
Not completed — Adverse Event | 13 | 5 | 2
Not completed — Withdrawal by Subject | 17 | 2 | 1
Not completed — Withdrawal by parent/guardian | 0 | 7 | 0
Not completed — Physician Decision | 2 | 1 | 1
Not completed — Lost to Follow-up | 2 | 1 | 0
Not completed — Lack of Efficacy | 2 | 0 | 1
Not completed — Other | 6 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety set: subjects who have received the investigational medicinal product (IMP) at least once
Groups:
- Total: Total of all reporting groups
Arm/Group | Adult: 1% OPA-15406 Ointment | Pediatric: 0.3% OPA-15406 Ointment | Pediatric: 1% OPA-15406 Ointment | Total
Number analyzed (Participants) | 166 | 144 | 56 | 366
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (11.3) | 7.1 (3.5) | 8.3 (3.5) | 7.4 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 63 | 18 | 146
  Male | 101 | 81 | 38 | 220
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 166 | 144 | 56 | 366
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 166 | 144 | 56 | 366

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Experiencing Treatment-Emergent Adverse Events (TEAEs)
Description: The number of subjects were calculated regarding adverse events occurring after IMP administration (=TEAEs).
Time Frame: Treatment period (52 weeks)
Population: Safety set: subjects who have received the IMP at least once
Measure: Count of Participants; unit: Participants
Arm/Group | Adult: 1% OPA-15406 Ointment | Pediatric: 0.3% OPA-15406 Ointment | Pediatric: 1% OPA-15406 Ointment
Number analyzed (Participants) | 166 | 144 | 56
Participants | 120 | 131 | 47

2. Secondary Outcome: Responder Rate of Investigator's Global Assessment (IGA)
Description: The investigator or subinvestigator assessed the skin symptoms using IGA. The investigator or subinvestigator scored the severity (0 = clear, 1 = almost clear, 2 =mild, 3 = moderate, 4 = severe/very severe) of the overall symptoms of the treatment area (erythema, infiltration, papules, effusion and scab formation) from baseline to Week 52.
  Incidence of success in IGA is defined as the rate of subjects whose IGA score is 0 (clear) or 1 (almost clear) and has improved by at least 2 grades (responders) from baseline.
Time Frame: Week 52
Population: Subjects who have received the IMP at least once and had IGA score at the baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adult: 1% OPA-15406 Ointment | Pediatric: 0.3% OPA-15406 Ointment | Pediatric: 1% OPA-15406 Ointment
Number analyzed (Participants) | 166 | 144 | 56
percentage of participants | 34.94 [27.71 to 42.71] | 52.78 [44.29 to 61.15] | 51.79 [38.03 to 65.34]

3. Secondary Outcome: Responder Rate of Eczema Area and Severity Index 75 (EASI 75)
Description: The investigator or sub investigator assessed the symptoms of AD using EASI. EASI's minimum and maximum scores are 0 and 72 scores respectively. The higher the EASI score is, the more severe the symptoms of AD. The investigator or sub investigator scored the severity (0-3 points) and affected body surface area (%) based on the 4 symptoms (erythema, infiltration/papules, excoriation, and lichenification) on the 4 body regions (face, neck and head ; upper limbs ;trunk; and lower limbs).
  EASI 75 is defined as the rate of subjects whose EASI score has improved at least 75% from baseline.
Time Frame: Week 52
Population: Subjects who have received the IMP at least once and had EASI score at the baseline.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adult: 1% OPA-15406 Ointment | Pediatric: 0.3% OPA-15406 Ointment | Pediatric: 1% OPA-15406 Ointment
Number analyzed (Participants) | 166 | 144 | 56
percentage of participants | 55.42 [47.52 to 63.13] | 77.08 [69.35 to 83.67] | 64.29 [50.36 to 76.64]

ADVERSE EVENTS:
Time Frame: Treatment period (52 weeks)
Description: Subjects who have received the IMP at least once were included in the safety analysis.
Arm/Group | Adult: 1% OPA-15406 Ointment | Pediatric: 0.3% OPA-15406 Ointment | Pediatric: 1% OPA-15406 Ointment
All-Cause Mortality (participants affected / at risk) | 0/166 | 0/144 | 0/56
Serious Adverse Events (participants affected / at risk) | 2/166 | 1/144 | 0/56
Other Adverse Events (participants affected / at risk) | 72/166 | 108/144 | 43/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult: 1% OPA-15406 Ointment (N=166) | Pediatric: 0.3% OPA-15406 Ointment (N=144) | Pediatric: 1% OPA-15406 Ointment (N=56)
Rhegmatogenous retinal detachment (Eye disorders) | 1 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adult: 1% OPA-15406 Ointment (N=166) | Pediatric: 0.3% OPA-15406 Ointment (N=144) | Pediatric: 1% OPA-15406 Ointment (N=56)
Conjunctivitis allergic (Eye disorders) | 5 | 14 | 7
Bronchitis (Infections and infestations) | 1 | 9 | 3
Folliculitis (Infections and infestations) | 10 | 9 | 5
Gastroenteritis (Infections and infestations) | 5 | 11 | 6
Impetigo (Infections and infestations) | 2 | 26 | 5
Influenza (Infections and infestations) | 5 | 21 | 4
Molluscum contagiosum (Infections and infestations) | 0 | 7 | 3
Nasopharyngitis (Infections and infestations) | 24 | 47 | 17
Pharyngitis (Infections and infestations) | 0 | 6 | 4
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 7 | 3
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 35 | 30 | 17
Dermatitis contact (Skin and subcutaneous tissue disorders) | 5 | 9 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 8 | 14 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-01): https://cdn.clinicaltrials.gov/large-docs/29/NCT03961529/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-23): https://cdn.clinicaltrials.gov/large-docs/29/NCT03961529/SAP_001.pdf